CLINICAL TRIAL: NCT02059473
Title: Treatment of Small Acute Full-thickness tears-a Prospective Randomised Controlled Trial
Brief Title: Treatment of Small Acute Cuff Tears, a Randomized Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Hanna Bjornsson, PHD, Orthopeadic shouldersurgeon, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: acutecufftearhannahallgren
Record Dates: First submitted 2014-02-04; First posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physiotherapy & Surgery (Experimental): Mini-open rotator cuff repair
  Interventions: Procedure: Rotator cuff repair; Procedure: Physiotherapy
- Physiotherapy (Active Comparator): Structured physiotherapy
  Interventions: Procedure: Physiotherapy

INTERVENTIONS:
Procedure: Rotator cuff repair — Physiotherapy & Surgery
  Arms: Physiotherapy & Surgery
Procedure: Physiotherapy

SUMMARY:
The purpose of this project is to compare operative repair of traumatically torn rotator cuff tendon with physiotherapy in a randomized prospective study.

DETAILED DESCRIPTION:
In clinical practice most patients with a traumatic acute rotator cuff tear are treated with operative repair. The results of surgery are in most cases good but there are also good results in the literature from conservative treatment. So far there has been no prospective randomized comparison between the two treatments. When it comes to degenerative non-traumatic tears, level 1 and 2 studies have not been able to show the superiority of surgery.

This study takes place in 2 clinics in Sweden (Linköping and Kalmar). Patients who have no previous shoulder conditions, a trauma to the shoulder and pain and/or inability to lift their arm will undergo magnetic resonance imaging (MRI). If this indicates a full-thickness rotator cuff tear of the cranial part of the rotator cuff the patient will be randomized to surgery or physiotherapy. Surgical intervention is mini-open repair.

Follow-up takes place at 3 months, 6 months and 12 months with patient scores taken by a blinded independent physiotherapist. At 12 months a new MRI is conducted as well.

ELIGIBILITY:
Inclusion Criteria:

* Trauma to the shoulder
* Full thickness cranial rotator cuff tear
* Operation possible within 3 months

Exclusion Criteria:

* 2 or more rotator cuff tendons involved
* Fracture
* Dislocation
* Previous shoulder condition (symptomatic osteoarthritis (Gleno-humeral (GH) joint, Acromial-Clavicular (AC) joint), frozen shoulder, instability, tumor)
* Malignancy
* Rheumatic disease
* Inability to understand swedish
* Substance abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley Shoulder Assessment score | Twelve months

SECONDARY OUTCOMES:
Western Ontario Rotator Cuff score | Twelve months
  Shoulder specific, patient reported outcome score
MRI | Twelve months
  Magnetic Resonance imaging. Gives a measure of muscle atrophy, fatty infiltration, rerupture and enlargement of the tendon rupture.

OTHER OUTCOMES:
Euro-Qol-five-Dimensions (EQ-5D) | Twelve months
  Quality of life assessment
Patient Global Impression of Change (PGIC) | Twelve months
  Patients Global impression of Change

CONTACTS AND LOCATIONS:
Overall Officials: Lars Adolfsson, Professor, Principal Investigator — Linkoeping University
Locations (1):
- Orthopedic Clinic, Linköping University Hospital, Linköping, Sweden